CLINICAL TRIAL: NCT02153437
Title: A Study of the Effects of BMS-919373 on Atrial Effective Refractory Period in Subjects With a Dual-Chamber Pacemaker
Brief Title: Study of the Effects of BMS-919373 on the Electrical Activity of the Heart Using Pacemakers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CV205-006
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Sotalol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: BMS-919373 (Experimental): BMS-919373 oral Solution/tablet single dose for one day
  Interventions: Drug: BMS-919373
- Arm B: Sotalol (Active Comparator): Sotalol oral Tablet single dose for one day
  Interventions: Drug: Sotalol
- Arm C: Placebo for BMS-919373 (Placebo Comparator): Oral solution/tablet one single dose for one day
  Interventions: Drug: Placebo for BMS-919373

INTERVENTIONS:
Drug: BMS-919373
  Other Names: iKUR
  Arms: Arm A: BMS-919373
Drug: Sotalol
  Other Names: Co Sotalol
  Arms: Arm B: Sotalol
Drug: Placebo for BMS-919373
  Arms: Arm C: Placebo for BMS-919373

SUMMARY:
To determine the effect of our compound (BMS-919373) on electrical activity of the heart using pacemakers.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria

* Age 18 years to 85 years.
* Eligible patients will have a dual-chamber permanent pacemaker.
* Women who are not of childbearing potential.

Exclusion Criteria

- Patients with a history of Atrial Fibrillation (AF) that is either:.

i) Permanent (i.e. patients are only in AF and never in sinus rhythm) or.

ii) Persistent (i.e. patients who's episodes of AF are longer than 7 days and require medical intervention, such as electrical or medical cardioversion, to return to sinus rhythm), are excluded.

* History of Transient Ischemic Attack (TIA) or stroke in the last 12 months.
* History of clinically significant ventricular arrhythmia (not including isolated monomorphic Premature Ventricular Contractions (PVCs)). Such arrhythmias are marked by loss of consciousness, emergent cardioversion or defibrillation or unstable vital signs requiring medical intervention.
* Complete heart block.
* Planned surgery, endovascular intervention or cardioversion within the study period.
* History of atrial fibrillation.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
The effect of BMS-919373 on Atrial effective refractory period (AERP) in subjects with a dual chamber pacemaker | At 0.5, 1, 2, and 4 hours following study drug administration

SECONDARY OUTCOMES:
The safety assessments will be based on Adverse event reports, vital sign measurements, Electrocardiogram (ECGs), physical examinations and clinical laboratory tests | At 1, 2, and 4 hours following study drug administration
Safety assessments based on Ventricular Effective Refractory Period (VERP) and change from baseline | At 2 hour following study drug administration
Safety assessments based on Atrioventricular interval (AVI) and change from baseline | At 1, 2, and 4 hours following study drug administration
Safety assessments based on Wenckebach cycle length (WCL) and change from baseline | At 1, 2, and 4 hours following study drug administration
Safety assessments based on Intra-atrial conduction time (IACT) and change from baseline | At 1, 2, and 4 hours following study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Local Institution, Austin, Texas, United States
- Canada (5):
  - The University Of Calgary, Calgary, Alberta
  - University Of Ottawa Heart Institute, Ottawa, Ontario
  - Local Institution - 0001, Toronto, Ontario
  - Local Institution - 0002, Montreal, Quebec
  - Local Institution, Montreal, Quebec

REFERENCES:
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html